CLINICAL TRIAL: NCT07184086
Title: The Effect of Cagrilintide and Semaglutide Combination Treatment Compared to a Weight-loss Inducing Diet on Energy Metabolism in Persons Living With Obesity: an Open-label Randomised Study
Brief Title: A Study to See How Metabolism is Influenced by Weight Loss Due to Intervention With Cagrilintide and Semaglutide Compared to Diet
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9838-8215; U1111-1316-8299 (Other: World Health Organization (WHO))
Record Dates: First submitted 2025-09-13; First posted 2025-09-19 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Caloric Restriction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CagriSema (Cagrilintide + Semaglutide) / CagriSema (Experimental): Participants will receive subcutaneous (s.c.) dose of CagriSema (cagrilintide B and semaglutide I) in a dose escalation regimen in Period A for up to 20 weeks and continue to receive the same dose escalation regimen until maximum dose is reached in Period B for up to 52 weeks.
  Interventions: Drug: CagriSema (Cagrilintide B + semaglutide I)
- Low Energy Diet (LED) / CagriSema (Experimental): Participants will receive a dietary intervention in period A for up to 20 weeks followed by a s.c. dose of CagriSema (cagrilintide B and semaglutide I) in a dose escalation regimen until maximum dose is reached in Period B for up to 52 weeks.
  Interventions: Drug: CagriSema (Cagrilintide B + semaglutide I); Behavioral: Low Energy Diet

INTERVENTIONS:
Drug: CagriSema (Cagrilintide B + semaglutide I) — Cagrilintide and semaglutide will be administered subcutaneously.
Behavioral: Low Energy Diet — Participants will receive dietary intervention as per diet intervention manual.
  Arms: Low Energy Diet (LED) / CagriSema

SUMMARY:
In this study we will be looking into how CagriSema influences metabolism (the process by which food is used to supply energy for the body) compared to a diet. CagriSema is a new investigational medicine. CagriSema cannot yet be prescribed by doctors but has previously been tested in humans. The study is split into 2 parts. In the first part of the study, participants will either get CagriSema or a weight loss diet (calorie reduced). In the second part of the study,all participants will get CagriSema. Which treatment participants get in the first part of the study is decided by chance. Like all medicines, the study medicine may have side effects. The study will last for about 1.5 years.

ELIGIBILITY:
Inclusion criteria:

* Male or female (sex assigned at birth).
* Age 18-65 years (both inclusive) at the time of signing the informed consent.
* Body Mass Index (BMI) greater than or equal to (≥) 30.0 kilograms per square meter (kg/m^2) at screening (Visit 1). Excess body weight should be due to excess adipose tissue, as judged by the investigator.

Exclusion criteria:

* Female who is pregnant, breast-feeding or intends to become pregnant or is of childbearing potential and not using highly effective contraceptive method.
* History of diabetes mellitus of any type, other than gestational diabetes mellitus.
* Claustrophobia or severe discomfort of being confined in small rooms.
* Contraindication for magnetic resonance imaging (MRI) scanning as per local guidance, including physical limitations that prevent the MRI scan.
* Unusual meal habits (including, but not limited to, eating disorders) and special diet requirements or unwillingness to eat the food provided in the study.
* Treatment with metformin or other glucose-lowering agent(s) within 90 days before screening (V1), regardless of indication.
* Treatment with any medication prescribed for the indication of obesity or weight management within 90 days before screening (Visit 1).
* Presence or history of malignant neoplasms or in situ carcinomas (other than basal or squamous cell skin cancer, low-risk prostate cancer, or in situ carcinomas of the cervix or carcinoma in situ/high grade prostatic intraepithelial neoplasia) within 5 years before screening (Visit 1).
* Physical measurement exceeding the dimensions or load capacity of the magnetic resonance imaging (MRI)/dual-energy X-ray absorptiometry (DEXA) scanner.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-26 (Actual); Primary Completion 2027-10-12 (Estimated); Study Completion 2027-10-12 (Estimated)

PRIMARY OUTCOMES:
Change in sleeping metabolic rate (SMR) | Baseline (Week 0) to Week 20
  Measured as kilojoules (kJ) per day.

SECONDARY OUTCOMES:
Change in 24-hour energy expenditure | Baseline (Week 0) to Week 20
  Measured as kJ per day.
Change in resting metabolic rate (RMR) | Baseline (Week 0) to Week 20
  Measured as kJ per day.
Change in basal metabolic rate (BMR) | Baseline (Week 0) to Week 20
  Measured as kJ per day.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (2):
- United States (2):
  - Advent Health-Res Inst, Orlando, Florida
  - Pennington Biomed Res Ctr, Baton Rouge, Louisiana

IPD SHARING:
Plan to Share IPD: Yes
According to the Novo Nordisk disclosure commitment on novonordisk-trials.com.
URL: https://novonordisk-trials.com